CLINICAL TRIAL: NCT05370547
Title: A Multiple Center Study on NOXA Expression-guided Randomized Chidamide Bridging Intervention in CAR-T Treated NHL Patients
Brief Title: Chidamide Bridging for CAR-T Therapy
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-071
Record Dates: First submitted 2022-05-07; First posted 2022-05-11 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Non Hodgkin's Lymphoma
Keywords: CAR-T; NOXA; Chidamide
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide; fludarabine; Cyclophosphamide; CF regimen; relmacabtagene autoleucel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- high NOXA expression (Experimental): NOXA IHC score > 4; Bridging therapy was allowed but not containing chidamide; n=60.
  Interventions: Drug: Fludarabine and cyclophosphamide; Biological: Anti-CD19 CAR-T cells
- low NOXA expression and no chidamide intervention (Experimental): NOXA IHC score < 4; Bridging therapy was allowed but not containing chidamide; n=30.
  Interventions: Drug: Fludarabine and cyclophosphamide; Biological: Anti-CD19 CAR-T cells
- low NOXA expression and chidamide intervention (Experimental): NOXA IHC score < 4; Bridging therapy containing chidamide alone or combination; n=30.
  Interventions: Drug: Chidamide; Drug: Fludarabine and cyclophosphamide; Biological: Anti-CD19 CAR-T cells

INTERVENTIONS:
Drug: Chidamide — 1. Chidamide monotherapy mode: Chidamide was administered for at least 6 times after leukapheresis, 10mg oral D1-4, 20mg oral D7 every 3 days to the beginning day of FC conditioning.
  2. Chidamide combination mode: The combination of one or more of the following drugs in addition to chidamide is permitted: glucocorticoids, BTK inhibitors, chemotherapy, other previously used resistance drugs, etc.
  Other Names: HDACi
  Arms: low NOXA expression and chidamide intervention
Drug: Fludarabine and cyclophosphamide — Patients should be received FC regimen conditioning 3 to 5 days prior to CAR-T cell infusion. The recommended regimen is intravenous fludarabine (25-30 mg/m^2) and cyclophosphamide (250-500 mg/m^2) daily for 3 consecutive days. The clinician may also adjust the cleansing regimen according to the patient's actual situation.
  Other Names: FC regimen
Biological: Anti-CD19 CAR-T cells — A single infusion of CAR-transduced autologous T cells administered intravenously at a target dose of 100 × 10^6 for Relma-cel or 2 × 10^6/kg for Axi-cel. Other commercial CAR-T doses are determined by specific drug infusion instructions. The dose of experimental CAR-T was determined by the investigator. Infusion volume was calculated based on CAR-T cell density and recommended dose.
  Other Names: Relma-cel; Axi-cel; Other commercial CAR-T cells; Experimental CAR-T cells

SUMMARY:
The previous research suggests that the low expression of NOXA protein may be an important biomarker for the treatment of drug resistance of chimeric antigen receptor-T (CAR-T) cells. Up regulating the expression of NOXA through histone deacetylase inhibitor (HDACi) can improve drug resistance and significantly improve the therapeutic effect of CAR-T cells. This study will enroll approximately 120 subjects with recurrent or refractory (r/r) B-cell non-Hodgkin's lymphoma (NHL). Those with high expression of NOXA will receive conventional CAR-T treatment (without chidamide bridging), and those with low expression of NOXA will be randomly assigned 1:1 to those without or containing chidamide bridging. The purpose of this study was to evaluate the clinical response and safety of chidamide bridging.

DETAILED DESCRIPTION:
Background:

CAR-T cell therapy has been shown to be superior to conventional therapy in patients with r/r B-cell NHL. However, prior clinical studies and real-world data suggest that approximately 30-40% of cases of drug resistance still occur after CAR-T cell therapy, and approximately 50-60% of cases have recurrent disease progression over time of infusion. The investigators used genome-wide CRISPR/Cas9 to screen for CAR T-resistant cells and identified low NOXA expression as associated with CAR-T resistance. NOXA protein is a member of the Bcl2 protein family, which plays a critical role in P53-dependent apoptosis. The previous research suggests that the low expression of NOXA protein may be an important biomarker for the treatment of drug resistance of CAR-T cells. Through the verification of nearly 40 clinical samples previously treated with CAR-T, the investigators found that low NOXA expression was associated with poor prognosis. Meanwhile, animal experiments demonstrated that HDACi can up-regulate the expression of NOXA in tumor cells and significantly improve the efficacy of CAR-T therapy by reducing the incidence of resistance. The research was published in Signal Transduction and Targeted Therapy in 2022.

Objective:

The primary objective of the study was to evaluate whether chidamide bridging intervention improved clinical response to CAR-T in patients with r/r B-cell NHL. A secondary objective was to evaluate the safety of bridging therapy with chidamide and subsequent CAR-T infusion in above patients. The exploratory objective was to investigate the effect of chidamide intervention on NOXA expression.

Design:

This is a multicenter, prospective, controlled, open-label, phase Ⅰ/Ⅱ study. 120 patients with r/r B-cell NHL will be enrolled. Biopsy was performed before peripheral blood mononuclear cell (PBMC) collection, and NOXA expression level was detected by immunohistochemistry (IHC).

Patients with high NOXA expression (IHC score > 4) were treated with conventional CAR-T process (n=60), including PBMC collection, bridging therapy (without chidamide), fludarabine and cyclophosphamide (FC) regimen conditioning, CAR-T cell infusion, efficacy evaluation and follow-up; Patients with low NOXA expression (IHC score 0 - 4) were randomly assigned 1:1 to conventional CAR-T group as mentioned earlier (n=30) or CAR-T group containing chidamide bridging therapy (n=30).

The bridging therapy regimen containing chidamide was divided into monotherapy and combination therapy. Chidamide combination intervention can be used in cases of high tumor burden, rapid progression of disease, symptoms of compression, involvement of specific sites or organs, and other burden reduction that need to be addressed. The combination of one or more of the following drugs in addition to chidamide is permitted: glucocorticoids, BTK inhibitors, chemotherapy, other previously used resistance drugs, etc.

In this study, commercial CAR-T cells (mainly Relma-cel, with Axi-cel or other commercial CAR-T cells also acceptable) or experimental CAR-T cells targeted at CD19 were acceptable.

If feasible, for the group with low NOXA expression, a secondary biopsy was performed at the same site to detect changes in NOXA expression before CAR-T infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Age 16-75, male or female;
2. Recurrent or refractory large B-cell lymphoma (LBCL) ,grade 1-3a follicular lymphoma (FL) and mantle cell lymphoma (MCL). Recurrent or refractory disease was defined as progression after systemic treatment with second-line or more lines (including CD20 monoclonal antibody and doxorubicin) or primary resistance (disease progression during first-line treatment or within 6 months after completion of treatment). LBCL includes diffuse large B-cell lymphoma non-specific type (DLBCL-NOS), diffuse large B-cell lymphoma transformed by follicular lymphoma (TFL), grade 3b FL, primary mediastinal large B-cell lymphoma (PMBCL), high-grade B-cell lymphoma with MYC and Bcl-2 and/or Bcl-6 rearrangement ( double strike/triple hit lymphoma, DHL/THL);
3. Eastern Cooperative Oncology Group (ECOG) physical status is 0-3;
4. Life expectancy ≥12 weeks;
5. Subjects must be willing to undergo either excised or large-needle lymph node or tissue biopsy, or provide lymph node or tissue biopsy from the most recent available archived tissue for immunohistochemical NOXA testing and pathology review in the study center laboratory;
6. There are measurable target lesions;
7. CD19 positive;
8. Are willing to use contraception according to the following criteria:

   A. Women of reproductive age (15-49 years) must undergo a pregnancy test with negative results within 7 days before starting treatment; B. Women of reproductive age should use effective contraception for at least 120 days after the last dose of the study drug (contraceptive success rate of at least 99%). The subject should communicate with the available contraceptive methods with at least 99% success rate and confirm the understanding of the period; C. Male subjects used effective contraception for at least 93 days after the last dose of study drug (contraceptive success rate of at least 99%). The subject should communicate with the available contraceptive methods with at least 99% success rate and confirm the understanding of the period; D. Infertile women (i.e., surgically sterilized by hysterectomy and/or bilateral oophorectomy or amenorrhea ≥12 months and age > 45 years) are not subject to conditions A and B above
9. Adequate bone marrow and organ functions (normal values shall not be obtained with growth factors, and hemocytopenia caused by lymphoma invasion of bone marrow is not subject to conditions A, B, and C below) :

A. Neutrophil count (ANC) ≥1.0×10^9/L; B. Hemoglobin ≥8.0g/dL; C. Platelet count ≥50×10^9/L; D. Total bilirubin ≤1.5× upper limit of normal value (ULN) (< 3 TIMES ULN for patients with Gilbert syndrome, cholestasis caused by hilar compression adenosis, biliary obstruction caused by liver involvement or lymphoma); E. Alanine aminotransferase/aspartate aminotransferase (ALT/AST) ≤2.5×ULN or ≤5×ULN when liver invasion is present; F. Creatinine clearance ≥40ml/min using the cockcroft-gault equation or glomerular filtration rate ≥40ml/min/1.73m2 using the modified renal disease diet formula; G. Lipase ≤1.5×ULN.

Exclusion Criteria:

1. Patients known to be allergic to the drug Chidamide;
2. Lymphoma involves the central nervous system;
3. Known human immunodeficiency virus (HIV) infection or immunopositive test;
4. Viral infections that cannot be controlled by antiviral drugs, such as herpetic virus infection, acute or chronic active hepatitis B, acute or chronic active hepatitis C, etc. [Note: chronic hepatitis B virus (HBV) carriers or non-active hepatitis B surface antigen (HBsAg) positive subjects and HBV-DNA lower than the detection limit can be included in the group; hepatitis C virus (HCV) antibody negative can be enrolled, HCV antibody positive patients need to be tested for HCV-RNA, if negative can be enrolled];
5. Presence of active infectious disease requiring treatment;
6. Received live vaccine within 30 days prior to enrollment;
7. Active autoimmune disease requiring systemic treatment within 12 months prior to enrollment (i.e., disease-modifying drugs, corticosteroids, or immunosuppressive drugs). Note: Alternative therapies (such as thyroxine, insulin, or physiologic corticosteroid replacement for adrenal or pituitary dysfunction) are not considered a systemic treatment;
8. History of severe allergic reactions;
9. Presence of congestive heart failure or uncontrolled arrhythmias classified by the New York Heart Association as class III-IV;
10. Patients with clinically significant electrocardiogram abnormalities and potential risk of malignant arrhythmias;
11. Clinically significant cardiac events, including unstable angina, acute myocardial infarction, and/or cardiac transmission problems, occurred within 6 months prior to enrollment;
12. A history of stroke or intracranial hemorrhage within 3 months prior to enrollment;
13. Major surgery or trauma occurred within 28 days prior to enrollment, or major side effects have not been recovered;
14. Accompanied by uncontrolled major medical conditions, including, but not limited to, kidney, liver, blood, gastrointestinal, endocrine, pulmonary, neurological, brain or psychiatric disorders;
15. Current or previous malignancy within 3 years prior to enrollment, excluding cured basal or squamous cell skin cancer, superficial bladder cancer, prostatic intraepithelial tumor and carcinoma in situ of the cervix;
16. Conditions in which a known mental or physical illness interferes with cooperation with the requirements of the study or disrupts the results or interpretation of the results and, in the opinion of the therapeutic investigator, makes the patient unfit for study participation;
17. There is the situation that the researcher's judgment will interfere with the whole study participation; Situations where there is significant risk to the subject; Or interferes with the interpretation of research data;
18. Pregnant or breast-feeding patients;
19. Inability to swallow and retain oral medications, malabsorption syndrome, diseases that significantly affect gastrointestinal function, total resection of the stomach or small intestine, ulcerative colitis, symptomatic inflammatory bowel disease, partial or complete intestinal obstruction;
20. Inability to understand or unwillingness to sign informed consent.

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants with progression-free survival (PFS) at 6 months after CAR-T infusion among all participants | 6 months
  PFS is defined as the time between the date of CAR-T infusion and disease progression or death from any cause. At the time of statistical analysis of study endpoints, there were no PFS events, and data were truncated as the date of the last objective tumor evaluation. Patients who were lost to follow-up or withdrew informed consent will be included in the end point evaluation, with data truncated as the date of the last objective tumor evaluation.

SECONDARY OUTCOMES:
Incidence of adverse events (AE) of chidamide bridging and subsequent CAR-T infusion arm | 12 months
  AE is defined as any adverse medical event from the time between the date of randomization and the date of 12 months after CAR-T infusion. AE may be an adverse sign (including abnormal laboratory tests, etc.), symptom, or illness that is not related to the purpose of medication and is time-related to drug use, regardless of causality to the drug, such as long-term cytopenia, cytokine release syndrome, neurotoxicity, etc.
Participants with objective response rate (ORR) at 3 months after CAR-T infusion among all participants | 3 months
  ORR was defined as the percentage of subjects who achieved complete response or partial response assessed by investigators and based on the Lugano 2014 assessment criterion. All subjects who do not meet objective response criteria by the data analysis deadline will be considered nonresponders. The source of this endpoint will only include the assessment of response obtained after CAR-T infusion and prior to any additional antitumor therapy.
Participants with complete response rate (CRR) at 3 months after CAR-T infusion among all participants | 3 months
  CRR was defined as the percentage of subjects who achieved a CR assessed by investigators and based on the Lugano 2014 assessment criterion.
Percentage of participants with recurrence-free survival (RFS) at 6 months after CAR-T infusion among all participants | 6 months
  RFS was defined as the time between the date of CAR-T infusion and the date of first lymphoma recurrence (local, regional, distant metastasis) or death (whatever the cause) for subjects who received complete response after CAR-T infusion. For participants who remained alive and whose disease had not recurred, RFS was censored on the date of last visit/contact with disease assessments.
Percentage of participants with RFS at 12 months after CAR-T infusion among all participants | 12 months
  RFS was defined as above.
Percentage of participants with PFS at 12 months after CAR-T infusion among all participants | 12 months
  PFS was defined as above.
Percentage of participants with overall survival (OS) at 12 months after CAR-T infusion among all participants | 12 months
  OS was defined as the time between the date of CAR-T infusion and death from any cause.

OTHER OUTCOMES:
Effect of chidamide intervention on NOXA expression | an average of 4 weeks
  For the group with low NOXA expression, a secondary biopsy was performed at the same site to detect changes in NOXA expression before CAR-T infusion. In the chidamide bridging group, the timing of secondary biopsy was arranged at least 6 times' chidamide therapy and before CAR-T infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, Ph.D, Principal Investigator — Biotherapeutic Department, Chinese PLA General Hospital
Locations (13):
- China (13):
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Peking University Cancer Hospital, Beijing, Beijing Municipality
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Sun Yat-Sen University Cancer Hospital, Guangzhou, Guangzhou
  - Tongji Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Xiehe Hospital, Tongji Medical College of HUST, Wuhan, Hubei
  - Tongji Hospital of Tongji University, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Soochow University, Suzhou, Suzhou
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
  - Biotherapeutic Department, Chinese PLA General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No